CLINICAL TRIAL: NCT07242989
Title: Outpatient Posterior Cervical Decompression, Instrumentation, and Fusion: The First Consecutive 100 Cases
Brief Title: Outpatient Posterior Cervical Fusion: Outcomes of the First 100 Consecutive Cases
Status: Completed | Type: Observational
Sponsor: NeuroSpine Center of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: TMW-2025-001
Record Dates: First submitted 2025-10-24; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cervical Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Posterior Cervical Decompression, Instrumentation and Fusion Patients: 100 consecutive patients with documented cervical spinal cord and/or nerve root compression unresponsive to conservative management.
  Interventions: Other: Enhanced recovery after surgery protocol

INTERVENTIONS:
Other: Enhanced recovery after surgery protocol — This is the only study evaluating OUTPATIENT posterior cervical decompression, instrumentation, and fusion patients in a prospective fashion with a median follow-up of 2.5 years.

SUMMARY:
Observational study regarding outcomes, complications, and patient acceptance for 100 consecutive patients undergoing outpatient posterior cervical decompression, instrumentation and fusion.

ELIGIBILITY:
Inclusion Criteria:

* patients with neurological signs and symptoms related to cervical stenosis, confirmed by MRI, who have failed to improve with appropriate conservative management.

Exclusion Criteria:

* patients who represent an inordinate risk to undergo general anesthesia in the outpatient setting.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult males and females referred to the NeuroSpine Center of Wisconsin in Appleton, WI, with cervical stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Neurologic Function (Modified JOA Score) | Baseline and 3 months post-operative
  Neurologic status will be assessed using the Modified Japanese Orthopaedic Association (mJOA) Score (1-18), with higher scores indicating better neurologic function.
Myelopathy Severity (Nurick Grade) | Baseline and 3 months post-operative
  Myelopathy severity will be measured using the Nurick Scale (Grades 0-5), with higher grades indicating greater impairment.
Pain Severity (VAS Neck and Arm Pain Scores) | Baseline, 3 months post-operative, and final follow-up (average 5 years)
  Pain will be assessed using the Visual Analog Scale (VAS) for neck and arm pain (0-10).
Functional Disability (Oswestry Neck Pain Index) | Baseline and 3 months post-operative
  Functional impairment will be assessed using the Oswestry Neck Pain Index (0-100%).
Surgical Outcome Rating (Odom Criteria) | 3 months post-operative and extended follow-up (average 5 years)
  Patient-reported surgical outcome will be graded using Odom Criteria (Excellent, Good, Fair, Poor).

SECONDARY OUTCOMES:
Number of Participants With Postoperative Complications or Readmissions | Day of surgery through study completion (average 5 years)
  All postoperative medical and surgical complications-including ER visits, unplanned admissions, and reoperations-will be recorded.
Number of Participants With Radiographic Evidence of Fusion or Hardware Failure | 6 weeks, 3 months, and extended follow-up (average 5 years)
  Radiographic evaluation of fusion status, hardware failure, and pseudoarthrosis will be performed using AP/lateral and flexion-extension cervical spine radiographs.

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroSpine Center of Wisconsin, Neenah, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT07242989/Prot_000.pdf